CLINICAL TRIAL: NCT01689337
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group, Phase II Trial to Investigate the Efficacy and Safety of 30 mcg and 100 mcg AS902330 Given as One Cycle of Three Intra-articular Knee Injections Once a Week for Three Weeks as an Adjunct Treatment to Patients Following Microfracture Surgery for Cartilage Injury of the Knee.
Brief Title: A Multicenter Trial of Sprifermin (AS902330 [Recombinant Human Fibroblast Growth Factor-18]) or Placebo After Microfracture Surgery for Cartilage Injury of the Knee
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was discontinued due to low recruitment.
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMR700692-007; 2012-001431-31 (EudraCT Number)
Record Dates: First submitted 2012-09-17; First posted 2012-09-21 (Estimated); Results first posted 2015-08-31 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Cartilage Injury of Knee
Keywords: Microfracture surgery; Cartilage repair; Knee surgery
MeSH Terms: interventions — fibroblast growth factor 18

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sprifermin (AS902330), 30 mcg (Experimental)
  Interventions: Drug: Sprifermin (AS902330)
- Sprifermin (AS902330), 100 mcg (Experimental)
  Interventions: Drug: Sprifermin (AS902330)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sprifermin (AS902330) — Sprifermin (AS902330) will be administered at a dose of 30 microgram (mcg) as intra-articular injection once every week for 3 weeks, starting from 2 weeks after MFx surgery.
  Arms: Sprifermin (AS902330), 30 mcg
Drug: Sprifermin (AS902330) — Sprifermin (AS902330) will be administered at a dose of 100 mcg as intra-articular injection once every week for 3 weeks, starting from 2 weeks after MFx surgery.
  Arms: Sprifermin (AS902330), 100 mcg
Drug: Placebo — Placebo matched to Sprifermin (AS902330) will be administered as intra-articular injection once every week for 3 weeks, starting from 2 weeks after MFx surgery.
  Arms: Placebo

SUMMARY:
This is a Phase 2, double-blind, multicenter, randomized, placebo-controlled trial to evaluate the efficacy and safety of Sprifermin (AS902330) (recombinant human fibroblast growth factor-18 [rhFGF-18]) as an adjunct treatment to subjects following microfracture (MFx) surgery for cartilage injury of the knee.

Primary Objectives

* To evaluate the effect of Sprifermin (AS902330) intra-articular knee injections as adjunct to microfracture (MFx) surgery on the composition of the refilled cartilage in the target knee, as measured by gadolinium-enhanced magnetic resonance imaging (MRI) of cartilage (dGEMRIC) time constant 1 (T1) relaxation time at 6 months after MFx surgery
* To evaluate the safety profile of Sprifermin (AS902330) when administered intra-articular into the knee as adjunct to MFx surgery in subjects with cartilage injury of the knee

Secondary Objectives

* To further support the efficacy and safety of Sprifermin (AS902330) as an adjunct to MFx for cartilage injury repair through symptomatic outcomes and quantitative MRI measurement

ELIGIBILITY:
Inclusion Criteria:

* Subjects with candidature for MFx surgery on the femoral articular surfaces (medial or lateral condyles or trochlear groove), with intact subchondral bone
* Subjects with moderate to severe pain in the target knee prior to surgery; average score greater than equal to (>=) 4.0 over 7 consecutive days on numeric rating scale of pain intensity (completed within 30 [+15] days before surgery)
* Intraoperative inclusion criteria: Subjects with 1 or 2 focal chondral lesions per target knee, where peripheral debridement to healthy cartilage results in all of the following:

  * Each lesion has an area of >= 1 square centimeter (cm^2) and less than equal to (<=) 4 cm^2
  * Each lesion is <= 6 millimeter (mm) in depth, as measured from the surrounding subchondral plate
  * Arthroscopic confirmation that each non-osteochondritis dissecans (OCD) lesion is between International Cartilage Repair Society (ICRS) Grades I and III (D); a Grade III non-OCD lesion is equivalent to an Outerbridge Grade IV lesion with minimal subchondral bone loss
* Other protocol-defined inclusion criteria could apply

Exclusion Criteria:

* Subjects with prior marrow stimulation treatment of the target knee, that is, MFx, micro-drilling, abrasion chondroplasty or cartilage repair including, but not limited to, autologous chondrocyte implantation (ACI), matrix/membrane autologous chondrocyte implantation (MACI), or osteochondral transplantation (autologous or allogeneic)
* Subjects with body mass index (BMI) of greater than 35 kilogram per square meter (kg/m^2) at screening
* Malalignment of the target knee greater than 5 degrees as measured from the mechanical axis, as confirmed by alignment (long bone) X-ray images
* Subjects with clinical and/or radiographic disease diagnosis of the target knee joint including, but not limited to the following: generalized osteoarthritis (OA), rheumatoid arthritis, or avascular necrosis
* Subjects who have any contraindication to MRI or gadolinium-based or iodinated contrast agents according to the site's standard practice guidelines
* Other protocol-defined exclusion criteria could apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2013-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono, Inc., Rockland MA, a subsidiary of Merck KGaA, Darmstadt, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sprifermin (AS902330) 30 microgram (mcg) and placebo arms were planned, but did not enroll participants due to early study discontinuation.
Groups:
- Sprifermin (AS902330), 100 mcg: Sprifermin (AS902330) was administered at a dose of 100 microgram (mcg) as intra-articular injection once every week for 3 weeks, starting from 2 weeks after microfracture (MFx) surgery.
Period: Overall Study
Arm/Group | Sprifermin (AS902330), 100 mcg
Started | 1
Completed | 0
Not Completed | 1
Not completed — Study Discontinuation | 1

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) analysis set included all participants randomly allocated to treatment.
Arm/Group | Sprifermin (AS902330), 100 mcg
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Gender [Count of Participants; unit: Participants]
  Female | 0
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Composition of the Refilled Cartilage Measured by Delayed Gadolinium-Enhanced Magnetic Resonance Imaging of Cartilage (dGEMRIC) Using T1 Relaxation Time at Month 6 Post-MFx Surgery
Description: The dGEMRIC is an imaging technique that estimates the proteoglycan (and glycosaminoglycan) content of joint cartilage using spin-lattice relaxation time T1 after penetration of gadolinium contrast agent. Composition of the refilled cartilage was to be reported.
Time Frame: 6 months post-MFx surgery
Population: Efficacy analysis was not performed as only one participant was enrolled in the study. The study was terminated due to low recruitment.
Groups:
- Sprifermin (AS902330), 100 mcg: Sprifermin (AS902330) was administered at a dose of 100 microgram (mcg) as intra-articular injection once every week for 3 weeks, starting from 2 weeks after MFx surgery.
Arm/Group | Sprifermin (AS902330), 100 mcg
Number analyzed (Participants) | 0

2. Secondary Outcome: Composition of the Refilled Cartilage Measured by dGEMRIC Using T1 Relaxation Time Beyond Month 6 Post-MFx Surgery
Description: as for outcome 1
Time Frame: Every 6 months up to 5 years beyond 6 months post-MFx surgery
Population: as for outcome 1
Arm/Group | Sprifermin (AS902330), 100 mcg
Number analyzed (Participants) | 0

3. Secondary Outcome: Change From Baseline in Participant-reported Outcome Measure: Knee Injury and Osteoarthritis Outcome Score (KOOS) Sub-scores for Pain and Activities of Daily Living (ADL)
Description: The KOOS Version LK1.0 is a knee-specific self-administered questionnaire used to assess pain, function, quality of life, and ADL. It consists of 42 items grouped into 5 subscales: pain, other symptoms (including swelling, restricted range of motion, and mechanical symptoms), function in ADL, function in sport and recreation (FSR), and impact on quality of life (QOL) (knee-related QOL, including awareness of the knee condition and changes in lifestyle). The subscales are scored separately; each yields a score between 0 and 100, with 0 representing extreme knee problems and 100 representing absence of problems. Total KOOS score is the average of all 5 subscale scores; ranging from 0 to 100; where 0 represents extreme knee problems and 100 represents absence of knee problems. Change from baseline in pain and ADL sub-scores was to be calculated by the respective scores at the specific time point minus the scores at baseline.
Time Frame: Every 6 months up to 5 years
Population: as for outcome 1
Arm/Group | Sprifermin (AS902330), 100 mcg
Number analyzed (Participants) | 0

4. Secondary Outcome: Change From Baseline in Participant-reported Outcome Measure: Total KOOS Score, Three KOOS Sub-scores and Total KOOS Minus FSR Sub-score
Description: The KOOS Version LK1.0 is a knee-specific self-administered questionnaire used to assess pain, function, quality of life, and ADL. It consists of 42 items grouped into 5 subscales: pain, other symptoms (including swelling, restricted range of motion, and mechanical symptoms), function in ADL, FSR, and impact on QOL (knee-related QOL, including awareness of the knee condition and changes in lifestyle). The subscales are scored separately; each yields a score between 0 and 100, with 0 representing extreme knee problems and 100 representing absence of problems. Total KOOS score is the average of all 5 subscale scores; ranging from 0 to 100; where 0 represents extreme knee problems and 100 represents absence of knee problems. Change from baseline in total KOOS score; other symptoms, knee-related QOL, and FSR sub-scores; and total KOOS minus FSR sub-score was to be calculated by the respective scores at the specific time point minus the scores at baseline.
Time Frame: Every 6 months up to 5 years
Population: as for outcome 1
Arm/Group | Sprifermin (AS902330), 100 mcg
Number analyzed (Participants) | 0

5. Secondary Outcome: Change From Baseline in Participant-reported Outcome Measure: Numeric Rating Scale (NRS) Score
Description: Knee pain was to be rated by the participant using an 11-point NRS of pain intensity. The NRS is scaled from 0 (no pain) to 10 (worst possible pain). Change from baseline in NRS score was to be calculated by the score at the specific time point minus the score at baseline.
Time Frame: Every 6 months up to 5 years
Population: as for outcome 1
Arm/Group | Sprifermin (AS902330), 100 mcg
Number analyzed (Participants) | 0

6. Secondary Outcome: Change From Baseline in Participant-reported Outcome Measure: Lower Extremity Activity Scale (LEAS) Score
Description: The LEAS is an 18-level single-question self-administered scale that has been validated as a clinical outcome measure for the assessment of participants' actual activity levels. The LEAS is scaled from 1 to 18, with 18 indicating levels of highest activity. Change from baseline in LEAS score was to be calculated by the score at the specific time point minus the score at baseline.
Time Frame: Every 6 months up to 5 years
Population: as for outcome 1
Groups:
- AS902330, 100 mcg: AS902330 was administered at a dose of 100 microgram (mcg) as intra-articular injection once every week for 3 weeks, starting from 2 weeks after MFx surgery.
Arm/Group | AS902330, 100 mcg
Number analyzed (Participants) | 0

7. Secondary Outcome: Change From Baseline in the Physician-reported Outcome Measure: Lysholm Knee Scale Score
Description: The Lysholm knee scale is a physician-reported outcome measure to assess knee function after ligament injury. It is scaled from 0 to 100 with higher scores representing better function. Change from baseline in Lysholm knee scale score was to be calculated by the score at the specific time point minus the score at baseline.
Time Frame: Every 6 months up to 5 years
Population: as for outcome 1
Arm/Group | Sprifermin (AS902330), 100 mcg
Number analyzed (Participants) | 0

8. Secondary Outcome: Composition of the Refilled Cartilage Using T2 Mapping
Description: The transverse relaxation time T2 mapping is an MRI technique that is able to evaluate collagen organization and orientation within cartilage. Composition of the refilled cartilage was to be reported.
Time Frame: Every 6 months up to 5 years
Population: as for outcome 1
Arm/Group | Sprifermin (AS902330), 100 mcg
Number analyzed (Participants) | 0

9. Secondary Outcome: Volume of the Refilled Cartilage
Description: Volume of the refilled cartilage was to be measured by MRI.
Time Frame: Every 6 months up to 5 years
Population: as for outcome 1
Arm/Group | Sprifermin (AS902330), 100 mcg
Number analyzed (Participants) | 0

10. Secondary Outcome: Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) Score
Description: The MOCART score is used to describe the constitution of the cartilage repair tissue and the surrounding structures.
Time Frame: Every 6 months up to 5 years
Population: as for outcome 1
Arm/Group | Sprifermin (AS902330), 100 mcg
Number analyzed (Participants) | 0

11. Secondary Outcome: Six-minute Walk Test
Description: Six (6)-minute walk test is used to measure gait function and for pre- and post-operative evaluation in cartilage injury repair. Maximum comfortable distance (in meters) that a participant can walk in 6 minutes was to be reported.
Time Frame: Every 3 months up to 5 years beyond Month 6 post-MFx surgery
Population: as for outcome 1
Arm/Group | Sprifermin (AS902330), 100 mcg
Number analyzed (Participants) | 0

12. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was defined as any new untoward medical occurrences/worsening of pre-existing medical condition without regard to possibility of causal relationship. An SAE is an AE that results in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect.
Time Frame: Baseline up to Month 60
Population: The safety analysis set included all participants who received at least 1 dose of trial drug.
Measure: Number; unit: participants
Arm/Group | Sprifermin (AS902330), 100 mcg
Number analyzed (Participants) | 1
participants
  Adverse Events | 1
  Serious Adverse Events | 0

ADVERSE EVENTS:
Time Frame: Up to 6 months
Description: An adverse event (AE) was defined as any new untoward medical occurrences/worsening of pre-existing medical condition, whether or not related to study drug.
Arm/Group | Sprifermin (AS902330), 100 mcg
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sprifermin (AS902330), 100 mcg (N=1)
Syncope (Nervous system disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Panic attack (Psychiatric disorders) | 1
Pyrexia (General disorders) | 1
Streptococcal pharyngitis (Infections and infestations) | 1
Knee swelling (Musculoskeletal and connective tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Efficacy analysis was not performed as only one participant was enrolled in the study. The study was terminated due to low recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor can with reasonable grounds require changes to the communication which do not change the scientific statement or neutrality of the communication.